CLINICAL TRIAL: NCT01017770
Title: Artemether-lumefantrine Vs Co-formulated Amodiaquine + Artesunate for the Treatment of Uncomplicated Falciparum Malaria: a Randomized Open-label Trial to Evaluate the Effectiveness of the Burkina Faso New Drug Policy
Brief Title: Artemether-lumefantrine (AL) Versus Artesunate + Amodiaquine (ASAQ) for the Treatment of Uncomplicated Falciparum Malaria in Burkina Faso
Acronym: ACTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Muraz (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Tinto Halidou, PharmD, PhD, Centre Muraz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTEffectiveness
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Uncomplicated P. Falciparum Malaria in Children
Keywords: Uncomplicated malaria
MeSH Terms: interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether -lumefantrine (Experimental): Experimental Treatment of malaria with Artemether-lumefantrine (AL), according to one of the two options given by national protocol in Burkina Faso
  Interventions: Drug: Artemether-lumefantrine
- Artesunate-amodiaquine (Experimental): Treatment of malaria with Artesunate-amodiaquine(AS-AQ), according to one of the two options given by national protocol in Burkina Faso
  Interventions: Drug: Artesunate-amodiaquine

INTERVENTIONS:
Drug: Artesunate-amodiaquine — Coformulated AQ+AS by Sanofi-Aventis has been pre-qualified by WHO in 2008. It is administered once daily for three consecutive days, and it is available in three different dosages (25mg/67.5mg; 50mg/135mg; 100mg/270mg)
  Other Names: ASAQ, Coarsucam
  Arms: Artesunate-amodiaquine
Drug: Artemether-lumefantrine — Artemether-lumefantrine by Novartis was the first fixed-dose ACT that was prequalified by WHO in April 2004. A 3-day, 6-dose regimen of AL is recommended for infants and children weighing 5-35 kg and adults weighing > 35 kg.
  Other Names: AL, Coartem(R), Riamet(R)
  Arms: Artemether -lumefantrine

SUMMARY:
Several countries in Africa have changed their first-line treatment for uncomplicated malaria to an ACT. Burkina Faso has changed its policy to Artemether-Lumefantrine (AL) and Artesunate-Amodiaquine (AQ+AS). However, such choice has been done without knowing the local effectiveness of these drugs when they are given to patients in real life conditions, without direct observation of the drug administration. Thus, this study aims at investigating the effectiveness of AQ+AS and AL, when given to children with uncomplicated malaria in Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 5 kg;
* Monoinfection with P. falciparum and a parasitaemia of 2,000-200,000 parasites /µl;
* Fever (axillary temperature ≥37.5 °C) or history of fever in the preceding 24 hours;
* Haemoglobin value above 5.0 g/dl;
* Absence of febrile conditions caused by diseases other than malaria.

Exclusion Criteria:

* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand;
* Signs of severe malaria (WHO 2000);
* Mixed malaria infection;
* Severe malnutrition;
* Other underlying diseases (cardiac, renal, hepatic diseases);
* History of allergy to study drugs;

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Polymerase chain reaction (PCR) adjusted treatment failure | Day 28

SECONDARY OUTCOMES:
Treatment failure up to day 42 (PCR adjusted and unadjusted) | Day 42
Gametocytes (prevalence and density) | At day 7, 14, 21, 28, 35 and 42 days after treatment
Hb changes | Day 35

CONTACTS AND LOCATIONS:
Locations (3):
- Burkina Faso (3):
  - Nanoro, Nanoro, Boulkiemdé
  - IRSS-DRO/Centre Muraz, Bobo-Dioulasso, Bp 545
  - Tinto Halidou, Bobo-Dioulasso, Houet